CLINICAL TRIAL: NCT02752750
Title: Longitudinal Quantitative Susceptibility Mapping (QSM) in Alzheimer 's Disease
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: QSM AD
Record Dates: First submitted 2016-04-19; First posted 2016-04-27 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- AD_GROUP: Patients with Alzheimer's disease
  Interventions: Other: MRI
- HC_GROUP: Healthy controls
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — MR imaging (MRI) at 3 Tesla
  Other Names: Magnetic resonance imaging

SUMMARY:
In this explorative longitudinal study 50 patients with Alzheimer's disease (AD) and 50 age-matched control subjects will be recruited for their 2 years follow-ups and undergo extensive cognitive testing and quantitative 3 Tesla magnetic resonance imaging (MRI). Regional differences of susceptibility and R2* relaxation rates in deep gray matter and the neocortex will be evaluated in AD patients and controls and related to the patients´ cognitive status at baseline.

DETAILED DESCRIPTION:
Abnormally increased brain iron accumulation in deep gray matter is a common finding in Alzheimer's disease (AD) and amyloid protein precursor and tau proteins were linked to disrupted iron homeostasis. Validation studies showed that brain iron can be measured precisely by the novel magnetic resonance imaging (MRI) technique quantitative susceptibility mapping (QSM) in vivo, thus, enabling reliable and precise longitudinal investigations.

It is hypothesized that pathologic brain iron accumulation can be assessed with higher sensitivity with QSM than with current MRI techniques such as R2* relaxation rate mapping and that regional QSM is a predictor for cognitive decline and disability.

This explorative longitudinal study is including 50 patients with AD and age-matched control subjects which will be recruited for their 2 years follow-ups and undergo extensive cognitive testing and quantitative 3 Tesla MRI. Regional differences of susceptibility and R2* in deep gray matter and the neocortex will be evaluated in AD patients and controls and related to the patients´ cognitive status at baseline. Follow-up MRI and clinical data with multivariate regression analysis serve to investigate the dynamics of AD-related changes of susceptibility, and their relation to cognitive functioning.

In conclusion, this explorative longitudinal study in a patient cohort aims to clarify whether regional QSM changes are potential biomarkers for AD progression.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of dementia according to DSM-IV and NINCDS-ADRDA criteria
* the patient lives either with the family or has less than 40h/week of external care
* the patients is able to understand the role in this study and is willing to participate
* the physician in charge of this study confirms that the patients understands the study and its aims according to cognitive and clinical testing

Exclusion Criteria:

* are other disorders
* participation in a clinical drug trial (phase 1-3)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Alzheimer 's Disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-05; Primary Completion 2024-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Quantitative magnetic susceptibility (QSM) in the human brain | 2 years
  Reveal the dynamics of disease related brain iron deposition (by QSM in ppm) and its relation to disease progression and cognition.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Langkammer, PhD, Principal Investigator — Medical University of Graz

IPD SHARING:
Plan to Share IPD: No